CLINICAL TRIAL: NCT05614284
Title: A Prospective, Post-Market, Multicenter Comparative Analysis of the Efficacy of Virtuos and Autograft Bone Graft in Lumbar Fusion Surgery
Brief Title: Comparative Analysis of Virtuos and Autograft in Lumbar Fusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol redesign.
Sponsor: Orthofix Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP - 2201VLF
Record Dates: First submitted 2022-11-04; First posted 2022-11-14 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Degenerative Disc Disease
Keywords: Lumbar Fusion; Cellular Based Lyograft; TLIF
MeSH Terms: conditions — Intervertebral Disc Degeneration | interventions — Transplantation, Autologous

STUDY DESIGN:
Intervention Model Description: 2:1 Enrollment: Virtuos vs. Autograft
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Virtuos (Experimental): Virtuos +/- Local Bone
  Interventions: Device: Virtuos
- Autograft (Active Comparator): Autograft +/- Allograft Chips
  Interventions: Device: Virtuos

INTERVENTIONS:
Device: Virtuos — Use of autograft or Virtuos Lyograft as an adjunct to spinal fusion in TLIF.
  Other Names: Autograft

SUMMARY:
Compare the lumbar fusion rates at 12 and 24 months when lumbar arthrodesis is performed using Virtuos or Autograft Bone Graft. Surgical approach is limited to TLIF (MIS or Open) with posterior fixation and supplemental posterolateral fusion as directed by physician, but must comply with FDA approved/cleared indication for use and labeling.

DETAILED DESCRIPTION:
The purpose of this study is to compare clinical and radiographic outcomes in patients undergoing transforaminal lumbar interbody fusion (minimally invasive or open) with either Virtuos bone graft or autograft/allograft bone graft.

Compare the lumbar fusion rates at 12 and 24 months when lumbar arthrodesis is performed using Virtuos or Autograft Bone Graft. Surgical approach is limited to TLIF (MIS or Open) with posterior fixation and supplemental posterolateral fusion as directed by physician, but must comply with FDA approved/cleared indication for use and labeling.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  1. At least 18 years of age at the time of surgery
  2. Undergoing lumbar spine fusion surgery with one of the following bone grafting options:

     1. Virtuos
     2. Virtuos with Autograft (local bone)
     3. Autograft
     4. Autograft + allograft (cancellous bone chips)
  3. Subject must have a documented diagnosis of DDD. DDD is defined by back and/or radicular pain with degeneration of the disc as confirmed by medical history, physical examination, and radiographic studies that may include CT, MRI, plain X-ray film, discography, myelography, etc. with one or more of the following findings:

     1. Instability as defined by >3mm translation or >5 degrees angulation
     2. Osteophyte formation of facet joints or vertebral endplates
     3. Decreased disc height, on average by >2mm, but dependent upon the spinal level
     4. Scarring/thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule
     5. Herniated nucleus pulposus
     6. Facet joint degeneration/changes; and/or
     7. Vacuum phenomenon
  4. Subject may have up to a Grade I Spondylolisthesis of the lumbar spine with clinical manifestations of one or more of the following phenomena:

     1. Radiculopathy
     2. Sensory deficit
     3. Motor weakness
     4. Reflex changes
  5. Subject must require lumbar posterolateral arthrodesis at 1-2 contiguous levels (L1-S1).
  6. The number of levels decompressed must equal the number of levels fused.
  7. Subject must have been unresponsive to conservative care for at least 6 months prior to fusion surgery.
  8. Subject must agree not to use electromagnetic adjuncts to enhance bone fusion during the course of the study
  9. Subject must be willing and able to sign an informed consent document.
  10. Subject must be willing and able to return for all follow-up visits, agree to participate in postoperative clinical and radiographic evaluations and comply with the required study regimen.

      Exclusion Criteria:

Exclusion criteria:

1. Subject is under 18 years of age (<18) at the time of consent
2. Subject has had prior lumbar spine fusion surgery at any level
3. Subject has greater than grade 1 spondylolisthesis of the lumbar spine
4. Subject is currently undergoing treatment for malignancy or has undergone treatment for malignancy in the past 5 years (benign skin cancer is permitted)
5. Subject is pregnant (confirmed by pregnancy test) or nursing or planning to become pregnant during the two years (24 months) following arthrodesis
6. Subject has an active local or systemic infection or is undergoing adjunctive treatment for local or systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-11-14 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Successful Fusion | Twelve months
  Fusion status at Twelve months postoperative

SECONDARY OUTCOMES:
Clinical Outcomes | Twelve months
  Patient Reported Outcomes (PROM): Disability and Pain
Safety Profile | Twelve and Twenty-four months
  Incidence of Adverse Events and Serious Adverse Events through Twelve and Twenty-four months.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Central CT Neurosurgery & Spine, New Britain, Connecticut
  - Michigan Brain and Spine, Royal Oak, Michigan
  - University of Texas South Western, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No